CLINICAL TRIAL: NCT01514279
Title: Targeting Obesity and Blood Pressure in Urban Youth(Consortium Title: Childhood Obesity Prevention and Treatment Research [COPTR] and Site Project Name IMPACT (Ideas Moving Parents and Adolescents to Change Together).
Brief Title: Ideas Moving Parents and Adolescents to Change Together (IMPACT)
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Elaine Borawski, Angela Bowen Williamson Professor of Community Nutrition, Director, Prevention Research Center for Healthy Neighborhoods, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMPACT-1-5U01HL103622-02; 5U01HL103622-02 (NIH)
Record Dates: First submitted 2011-12-20; First posted 2012-01-23 (Estimated); Results first posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Overweight; Obese
Keywords: Overweight; Obese; Over Nutrition; Nutrition Disorders; Body weight; Signs and Symptoms
MeSH Terms: conditions — Overweight; Obesity; Nutrition Disorders; Body Weight; Signs and Symptoms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HealthyCHANGE (Experimental): Cognitive behavioral strategies to address diet, physical activity, sedentary behavior and sleep for children.
  Interventions: Behavioral: HealthyCHANGE
- SystemCHANGE (Experimental): Intervention (based on systems improvement and choice architecture theories) System improvement and choice architecture theories seek to teach a set of skills using family self-designed experiments to redesign daily routines
  Interventions: Behavioral: SystemCHANGE
- Tools4CHANGE (No Intervention): In contrast to the behavioral arms, youths with their parent(s)/guardian randomized to this group will have one 60-minute face-to-face meeting at initiation of the study with a dietitian who is also trained in recommendations for exercise and sedentary behavior.

INTERVENTIONS:
Behavioral: HealthyCHANGE — Cognitive behavioral strategies to address diet, physical activity, sedentary behavior and sleep for children.
  It involves an intensive series of group sessions, followed by rotating monthly face-to-face meetings or phone calls.
  Arms: HealthyCHANGE
Behavioral: SystemCHANGE — Intervention (based on systems improvement and choice architecture theories) System improvement and choice architecture theories seek to teach a set of skills using family self-designed experiments to redesign daily routines regarding eating, activity and sleep.
  It involves an intensive series of group sessions, followed by rotating monthly face-to-face meetings or phone calls.
  Arms: SystemCHANGE

SUMMARY:
The National Heart, Lung, and Blood Institute (NHLBI) of the National Institute of Health (NIH) has sponsored a consortium of four sites across the United States, entitled Childhood Obesity Prevention and Treatment Research (COPTR). Each site has its own protocol. Case Western Reserve/Cleveland's project is entitled "Targeting Obesity and Blood Pressure in Urban Youth". The site name is IMPACT (Ideas Moving Parents and Adolescents to Change Together).

The project assesses the effects of three interventions on Body Mass Index(BMI) in overweight and obese urban 5th-8th grade youth: a cognitive-behavioral intervention (HealthyChange), a systems improvement intervention (SystemsChange), and an education-only intervention (Tools4Change). In addition the study assesses the potential additional impact of a school-community based intervention on outcomes.

The project has two phases: a formative phase (including focus groups and a pilot) and the main trial. The main trial will take place over approximately four years.

DETAILED DESCRIPTION:
The IMPACT trial will involve a 3-arm randomized controlled trial of three behavioral and educational interventions: (1) HealthyCHANGE, a behavioral approach focusing on building skills and increasing intrinsic motivation (based on cognitive-behavioral theory with motivational interviewing components); (2) SystemCHANGE, an innovative behavioral approach focusing on system re-design of the family environment and daily routines (based on social-ecological and personal process improvement theories); and (3) education-only (representing usual care, called Tools4CHANGE).

In the main trial, approximately half of the children will also be in schools that take part in the We Run This City (WRTC)Marathon program, a school-based fitness program administered by the YMCA, and half will be in schools that do not take part in the WRTC program.

This study will assess the impact of the interventions on the main trial's (1) primary outcome, Change in Body Mass Index (BMI). (2) secondary outcomes including diet, physical activity, sedentary behavior, sleep, blood pressure, cardiovascular risk, body composition, fitness, and quality of life (3) mediators including : child's self-efficacy, social support, motivation, family problem solving ability, systems thinking, and self-regulation;(4) moderators including: socioeconomic status, demographic factors, environmental factors, personal and psychosocial characteristics of child and parent.

ELIGIBILITY:
Inclusion Criteria:

* Students entering the 6th grade who are found at the standard school screenings to be overweight or obese
* (BMI 85th- 94th percentile or > 95th percentile for age/sex respectively)

Exclusion Criteria:

* Taking medications that alter appetite or weight (e.g. glucocorticoids, metformin, insulin, Risperidone (Risperdal), Olanzapine (Zyprexa), Clozapine(Clozaril), Quetiapine (Seroquel), Ziprasidone (Geodon), Carbamazepine (Tegretol), Valproic acid (Depakote/Depakene/Depacon), Aripiprazole (Abilify), Orlistat (Xenical), Sibutramine (Meridia), Phentermine, Diethylproprion (Tenuate), Topirimate (Topamax), glitazones (thiazolidinediones)
* Inability to understand English
* Stage 2 hypertension or stage 1 hypertension with end organ damage (left ventricular hypertrophy, microalbuminuria)
* Severe behavioral problems that preclude group participation (as reported by parent/guardian)
* Child involvement in another weight management program
* Family expectation to move from the region within 1 year
* The presence of a known medical condition that itself causes obesity (e.g., Prader-Willi syndrome) or interfere with HbA1C ( sickle cell disease)

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2011-02-01 (Actual); Primary Completion 2017-01-21 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine A Borawski, PhD, Principal Investigator — Case Western Reserve University; Shirley M Moore, RN, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Conducted in conjunction with the Research Coordinating Unit (UNC Chapel Hill) of the COPTR Consortium.

REFERENCES:
- [Background] Moore SM, Borawski EA, Cuttler L, Ievers-Landis CE, Love TE. IMPACT: a multi-level family and school intervention targeting obesity in urban youth. Contemp Clin Trials. 2013 Nov;36(2):574-86. doi: 10.1016/j.cct.2013.08.009. Epub 2013 Sep 2. PMID 24008055
- [Derived] Schuler BR, Gardenhire RA, Jones SD, Spilsbury JC, Moore SM, Borawski EA. Exploring the Association Between Trauma, Instability, and Youth Cardiometabolic Health Outcomes Over Three Years. J Adolesc Health. 2024 Feb;74(2):301-311. doi: 10.1016/j.jadohealth.2023.08.049. Epub 2023 Oct 15. PMID 37843478
- [Derived] JaKa MM, Wood C, Veblen-Mortenson S, Moore SM, Matheson D, Stevens J, Atkins L, Michie S, Adegbite-Adeniyi C, Olayinka O, Po'e EK, Kelly AM, Nicastro H, Bangdiwala SI, Barkin SL, Pratt C, Robinson TN, Sherwood NE. Applying the Behavior Change Technique Taxonomy to Four Multicomponent Childhood Obesity Interventions. West J Nurs Res. 2021 May;43(5):468-477. doi: 10.1177/0193945920954782. Epub 2020 Sep 10. PMID 32909523
- [Derived] Truesdale KP, Matheson DM, JaKa MM, McAleer S, Sommer EC, Pratt CA. Baseline diet quality of predominantly minority children and adolescents from households characterized by low socioeconomic status in the Childhood Obesity Prevention and Treatment Research (COPTR) Consortium. BMC Nutr. 2019 Sep 9;5:38. doi: 10.1186/s40795-019-0302-y. eCollection 2019. PMID 32153951
- [Derived] Cui Z, Truesdale KP, Robinson TN, Pemberton V, French SA, Escarfuller J, Casey TL, Hotop AM, Matheson D, Pratt CA, Lotas LJ, Po'e E, Andrisin S, Ward DS. Recruitment strategies for predominantly low-income, multi-racial/ethnic children and parents to 3-year community-based intervention trials: Childhood Obesity Prevention and Treatment Research (COPTR) Consortium. Trials. 2019 May 28;20(1):296. doi: 10.1186/s13063-019-3418-0. PMID 31138278
- [Derived] Moore SM, Borawski EA, Love TE, Jones S, Casey T, McAleer S, Thomas C, Adegbite-Adeniyi C, Uli NK, Hardin HK, Trapl ES, Plow M, Stevens J, Truesdale KP, Pratt CA, Long M, Nevar A. Two Family Interventions to Reduce BMI in Low-Income Urban Youth: A Randomized Trial. Pediatrics. 2019 Jun;143(6):e20182185. doi: 10.1542/peds.2018-2185. PMID 31126971

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between May 2012 and January 2014 as part of an existing BMI and blood pressure screening program in the local school district. Participants were randomly assigned to 1 of 3 intervention study arms within 37 days of the baseline clinical visit once recruited.
Groups:
- HealthyCHANGE: Cognitive behavioral strategies to address diet, physical activity, sedentary behavior and sleep for children.
  HealthyCHANGE: Cognitive behavioral strategies to address diet, physical activity, sedentary behavior and sleep for children.
  It involves an intensive series of group sessions, followed by rotating monthly face-to-face meetings or phone calls.
- SystemCHANGE: Intervention (based on systems improvement and choice architecture theories) System improvement and choice architecture theories seek to teach a set of skills using family self-designed experiments to redesign daily routines
  SystemCHANGE: Intervention (based on systems improvement and choice architecture theories) System improvement and choice architecture theories seek to teach a set of skills using family self-designed experiments to redesign daily routines regarding eating, activity and sleep.
  It involves an intensive series of group sessions, followed by rotating monthly face-to-face meetings or phone calls.
Period: Overall Study
Arm/Group | HealthyCHANGE | SystemCHANGE | Tools4CHANGE
Started | 118 | 123 | 119
Completed | 107 | 110 | 114
Not Completed | 11 | 13 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HealthyCHANGE | SystemCHANGE | Tools4CHANGE | Total
Number analyzed (Participants) | 118 | 123 | 119 | 360
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.58 (0.56) | 11.59 (0.59) | 11.51 (0.56) | 11.56 (0.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 73 | 69 | 208
  Male | 52 | 50 | 50 | 152
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Child's Race/Ethnicity: Non-Hispanic White | 4 | 5 | 5 | 14
  Child's Race/Ethnicity: Non-Hispanic Black | 91 | 92 | 93 | 276
  Child's Race/Ethnicity: Hispanic | 17 | 24 | 18 | 59
  Child's Race/Ethnicity: Multi-racial | 5 | 1 | 2 | 8
  Child's Race/Ethnicity: Other | 1 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 118 | 123 | 119 | 360
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 27.25 (4.78) | 27.36 (5.12) | 26.80 (4.71) | 27.14 (4.87)

OUTCOME MEASURES:

1. Primary Outcome: Slope of Body Mass Index (BMI)
Description: BMI slope (trajectory over 3 years) was created for each participant with outcomes multiply imputed for children without BMI values post-baseline. An F test with two numerator degrees of freedom was used to test for between-group differences using an alpha of .05.
Time Frame: Baseline, 12 mos, 24 mos and 36 mos
Measure: Mean (Standard Deviation); unit: kg/m^2/year
Arm/Group | HealthyCHANGE | SystemCHANGE | Tools4CHANGE
Number analyzed (Participants) | 112 | 117 | 117
kg/m^2/year | 0.821 (1.363) | 1.083 (1.129) | 0.952 (1.318)

2. Secondary Outcome: Dietary Intake- Calories Per Day
Description: Annualized change in calories per day.
  Dietary intake slopes (trajectory over 3 years) were created for each participant with outcomes multiply imputed for children without diet recall data post-baseline. An F test with two numerator degrees of freedom was used to test for between-group differences using an alpha of .05.
Time Frame: Baseline, 12 mos, 24 mos and 36 mos
Measure: Mean (Standard Deviation); unit: kcal/d/year
Arm/Group | HealthyCHANGE | SystemCHANGE | Tools4CHANGE
Number analyzed (Participants) | 106 | 113 | 116
kcal/d/year | 12.49 (226.65) | 6.99 (211.04) | 24.03 (250.44)

3. Secondary Outcome: Blood Pressure
Description: Annualized change in blood pressure measures using the slope of 3 year trajectory.
  Blood pressure slopes (trajectory over 3 years) were created for each participant with outcomes multiply imputed for children without blood pressure readings post-baseline. An F test with two numerator degrees of freedom was used to test for between-group differences using an alpha of .05.
Time Frame: Baseline, 12 mos, 24 mos and 36 mos
Measure: Mean (Standard Deviation); unit: mmHg/year
Arm/Group | HealthyCHANGE | SystemCHANGE | Tools4CHANGE
Number analyzed (Participants) | 112 | 116 | 117
mmHg/year
  Systolic Blood Pressure | 1.245 (3.319) | 1.130 (3.075) | 0.886 (2.787)
  Diastolic Blood Pressure | -0.136 (2.796) | -0.074 (2.726) | -0.162 (2.378)
  Systolic Blood Pressure Percentile | -1.450 (9.206) | -2.044 (8.063) | -2.028 (8.095)
  Diastolic Blood Pressure Percentile | -2.335 (8.228) | -2.044 (8.063) | -2.132 (6.645)

4. Secondary Outcome: Physical Activity
Description: Annualized change in physical activity measures of moderate to vigorous minutes per day and bed rest/sedentary minutes per day as measured by accelerometer.
  Physical activity slopes (trajectory over 3 years) were created for each participant with outcomes multiply imputed for children without accelerometer readings post-baseline. An F test with two numerator degrees of freedom was used to test for between-group differences using an alpha of .05.
Time Frame: [Baseline, 12 mos, 24 mos and 36 mos]
Measure: Mean (Standard Deviation); unit: minutes/day/year
Arm/Group | HealthyCHANGE | SystemCHANGE | Tools4CHANGE
Number analyzed (Participants) | 101 | 105 | 109
minutes/day/year
  Number of moderate/vigorous minutes per day | -3.370 (10.123) | -4.619 (7.486) | -3.523 (8.493)
  Number of bed rest/sedentary minutes per day | 10.501 (16.365) | 13.052 (14.561) | 11.022 (16.961)

5. Secondary Outcome: Sleep
Description: The results reflect the annualized change in adolescent sleep wake scale and pediatric daytime sleepiness scale. The items of the adolescent sleep wake scale are recoded to have a minimum of 0 and maximum value of 5, in which a higher scores for both the individual items and the overall sum score indicate a better outcome. The items of the pediatric daytime sleepiness are recoded to have a minimum of 0 and maximum value of 4, in which a lower score for both the individual items and the overall sum score indicates a better outcome.
  Sleep slopes (trajectory over 3 years) were created for each participant with outcomes multiply imputed for children without post-baseline measures. An F test with two numerator degrees of freedom was used to test for between-group differences using an alpha of .05.
Time Frame: [Baseline, 12 mos, 24 mos and 36 mos]
Measure: Mean (Standard Deviation); unit: score on a scale/year
Arm/Group | HealthyCHANGE | SystemCHANGE | Tools4CHANGE
Number analyzed (Participants) | 111 | 115 | 117
score on a scale/year
  Adolescent Sleep Wake | -1.061 (8.937) | -1.552 (9.755) | -1.184 (7.749)
  Pediatric Daytime Sleepiness | -0.239 (2.350) | -0.361 (2.618) | -0.273 (2.089)

6. Secondary Outcome: Cardiometabolic Factors- Fasting Glucose, HDL Cholesterol, LDL Cholesterol, Total Cholesterol
Description: Annualized change in various cardiometabolic factor measures over 3 years.
  Cardiometabolic factor slopes (trajectory over 3 years) were created for each participant with outcomes multiply imputed for children without blood draws post-baseline. An F test with two numerator degrees of freedom was used to test for between-group differences using an alpha of .05.
  Change in the slopes of fasting glucose, HDL cholesterol, LDL cholesterol, and total cholesterol over 3 years reported.
Time Frame: Baseline, 12 mos, 24 mos and 36 mos
Measure: Mean (Standard Deviation); unit: mg/dL/year
Arm/Group | HealthyCHANGE | SystemCHANGE | Tools4CHANGE
Number analyzed (Participants) | 102 | 106 | 108
mg/dL/year
  Fasting glucose | -0.146 (2.864) | -0.520 (3.805) | -0490 (3.135)
  HDL cholesterol | -0.300 (3.433) | -0.600 (2.526) | -0.385 (2.906)
  LDL cholesterol | -1.449 (7.915) | -1.970 (7.295) | -2.357 (6.645)
  Total cholesterol | -2.409 (9.500) | -3.651 (8.280) | -2.94 (7.201)

7. Secondary Outcome: Body Composition- BMI Percentile
Description: The annualized change in body composition measures over 3 years.
  Body composition slopes (trajectory over 3 years) were created for each participant with outcomes multiply imputed for children without body composition measurements post-baseline. An F test with two numerator degrees of freedom was used to test for between-group differences using an alpha of .05.
  Change in slope of BMI percentile over time reported.
Time Frame: Baseline, 12 mos, 24 mos and 36 mos
Measure: Mean (Standard Deviation); unit: BMI percentile/year
Arm/Group | HealthyCHANGE | SystemCHANGE | Tools4CHANGE
Number analyzed (Participants) | 109 | 114 | 114
BMI percentile/year | -1.375 (3.821) | -0.258 (1.552) | -1.082 (3.225)

8. Secondary Outcome: Fitness
Description: The annualized change in pacer laps completed during PACER test over 3 years.
  PACER test slopes (trajectory over 3 years) were created for each participant with outcomes multiply imputed for children without PACER test measurements post-baseline. An F test with two numerator degrees of freedom was used to test for between-group differences using an alpha of .05.
Time Frame: Baseline, 12 mos, 24 mos and 36 mos
Measure: Mean (Standard Deviation); unit: laps completed/year
Arm/Group | HealthyCHANGE | SystemCHANGE | Tools4CHANGE
Number analyzed (Participants) | 106 | 109 | 109
laps completed/year | 1.084 (2.640) | 0.533 (3.663) | 1.715 (3.491)

9. Secondary Outcome: Quality of Life- Perceived Stress
Description: The annualized change in perceived stress over 3 years. Participants are asked to rate individual scale items on their perception of how often they feel specific stressors on a scale from 0 (never) to 4 (very often). Individual scale items are summed for a total score. Higher scores indicate higher perceived frequency of stressors, therefore higher perceived stress. Outcomes are reported as the mean of the slope estimates for total perceived stress score over 3 years (from baseline to 36 months).
  The perceived stress slope (trajectory over 3 years) was created for each participant with outcomes multiply imputed for children without stress scores post-baseline. An F test with two numerator degrees of freedom was used to test for between-group differences using an alpha of .05.
Time Frame: [Baseline, 12 mos, 24 mos and 36 mos]
Measure: Mean (Standard Deviation); unit: scores on a scale/year
Arm/Group | HealthyCHANGE | SystemCHANGE | Tools4CHANGE
Number analyzed (Participants) | 109 | 115 | 117
scores on a scale/year | 0.313 (2.620) | -0.049 (2.769) | -0.026 (2.491)

10. Secondary Outcome: Dietary Intake- Percent Calories From Fat
Description: The annualized change of percent of calories from fat over 3 years.
  Percent calories from fat slope (trajectory over 3 years) was created for each participant with outcomes multiply imputed for children without diet recall data post-baseline. An F test with two numerator degrees of freedom was used to test for between-group differences using an alpha of .05.
Time Frame: Baseline, 12 months, 24 months, 36 months
Measure: Mean (Standard Deviation); unit: percent/year
Arm/Group | HealthyCHANGE | SystemCHANGE | Tools4CHANGE
Number analyzed (Participants) | 106 | 113 | 116
percent/year | 0.139 (2.905) | -0.050 (2.589) | -0.055 (0.360)

11. Secondary Outcome: Dietary Intake- Fruit and Vegetable Servings
Description: The annualized change in the number of fruit and vegetable servings per day over 3 years.
  Serving slopes (trajectory over 3 years) were created for each participant with outcomes multiply imputed for children without diet recall data post-baseline. An F test with two numerator degrees of freedom was used to test for between-group differences using an alpha of .05.
Time Frame: Baseline, 12 months, 24 months, 36 months
Measure: Mean (Standard Deviation); unit: number of servings/day/year
Arm/Group | HealthyCHANGE | SystemCHANGE | Tools4CHANGE
Number analyzed (Participants) | 106 | 113 | 116
number of servings/day/year
  Number of fruit servings per day | -0.061 (0.239) | -0.050 (0.234) | -0.055 (0.360)
  Number of vegetable servings per day | 0.013 (0.276) | 0.008 (0.263) | -0.008 (0.253)

12. Secondary Outcome: Dietary Intake- Sodium
Description: The annualized change in sodium intake (mg) per day over 3 years.
  Sodium intake slope (trajectory over 3 years) was created for each participant with outcomes multiply imputed for children without diet recall data post-baseline. An F test with two numerator degrees of freedom was used to test for between-group differences using an alpha of .05.
Time Frame: Baseline, 12 months, 24 months, 36 months
Measure: Mean (Standard Deviation); unit: mg/day/year
Arm/Group | HealthyCHANGE | SystemCHANGE | Tools4CHANGE
Number analyzed (Participants) | 106 | 113 | 116
mg/day/year | -0.42 (425.79) | 26.46 (409.34) | 39.15 (446.28)

13. Secondary Outcome: Cardiometabolic Factors- Hemoglobin A1c
Description: Annualized change in various cardiometabolic factor measures over 3 years.
  Cardiometabolic factor slopes (trajectory over 3 years) were created for each participant with outcomes multiply imputed for children without blood draws post-baseline. An F test with two numerator degrees of freedom was used to test for between-group differences using an alpha of .05.
  Change in the slope of glycated Hemoglobin A1c over 3 years reported.
Time Frame: [Baseline, 12 mos, 24 mos, 36 mos]
Measure: Mean (Standard Deviation); unit: % glycated/year
Arm/Group | HealthyCHANGE | SystemCHANGE | Tools4CHANGE
Number analyzed (Participants) | 102 | 106 | 108
% glycated/year | -0.040 (0.210) | -0.021 (0.304) | -0.017 (0.093)

14. Secondary Outcome: Cardiometabolic Factors- High-sensitivity C-reactive Protein
Description: Annualized change in various cardiometabolic factor measures over 3 years.
  Cardiometabolic factor slopes (trajectory over 3 years) were created for each participant with outcomes multiply imputed for children without blood draws post-baseline. An F test with two numerator degrees of freedom was used to test for between-group differences using an alpha of .05.
  Change in the slope of high-sensitivity C-reactive protein over 3 years reported.
Time Frame: [Baseline, 12 mos, 24 mos, 36 mos]
Measure: Mean (Standard Deviation); unit: mg/L/year
Arm/Group | HealthyCHANGE | SystemCHANGE | Tools4CHANGE
Number analyzed (Participants) | 102 | 106 | 108
mg/L/year | -0.013 (0.163) | -0.002 (0.141) | -0.0185 (0.123)

15. Secondary Outcome: Cardiometabolic Factors- Insulin
Description: Annualized change in various cardiometabolic factor measures over 3 years.
  Cardiometabolic factor slopes (trajectory over 3 years) were created for each participant with outcomes multiply imputed for children without blood draws post-baseline. An F test with two numerator degrees of freedom was used to test for between-group differences using an alpha of .05.
  Change in the slope of insulin over 3 years reported.
Time Frame: [Baseline, 12 mos, 24 mos, 36 mos]
Measure: Mean (Standard Deviation); unit: uU/mL/year
Arm/Group | HealthyCHANGE | SystemCHANGE | Tools4CHANGE
Number analyzed (Participants) | 102 | 106 | 108
uU/mL/year | 0.772 (4.761) | 0.406 (6.875) | 0.228 (4.568)

16. Secondary Outcome: Cardiometabolic Factors- HOMA-IR
Description: Annualized change in various cardiometabolic factor measures over 3 years.
  Cardiometabolic factor slopes (trajectory over 3 years) were created for each participant with outcomes multiply imputed for children without blood draws post-baseline. An F test with two numerator degrees of freedom was used to test for between-group differences using an alpha of .05.
  Change in the slope of HOMA-IR over 3 years reported.
Time Frame: [Baseline, 12 mos, 24 mos, 36 mos]
Measure: Mean (Standard Deviation); unit: score on a scale/year
Arm/Group | HealthyCHANGE | SystemCHANGE | Tools4CHANGE
Number analyzed (Participants) | 102 | 106 | 108
score on a scale/year | 0.032 (1.003) | 0.037 (1.281) | 0.004 (1.009)

17. Secondary Outcome: Body Composition- Waist-to-height Ratio
Description: The annualized change in body composition measures over 3 years.
  Body composition slopes (trajectory over 3 years) were created for each participant with outcomes multiply imputed for children without body composition measurements post-baseline. An F test with two numerator degrees of freedom was used to test for between-group differences using an alpha of .05.
  Change in slope of waist-to-height ratio over time reported. The weight-to-heigh ratio compares the child's waist circumference (cm) to their height (cm).
Time Frame: [Baseline, 12 mos, 24 mos, 36 mos]
Measure: Mean (Standard Deviation); unit: ratio/year
Arm/Group | HealthyCHANGE | SystemCHANGE | Tools4CHANGE
Number analyzed (Participants) | 109 | 114 | 114
ratio/year | -0.003 (0.023) | 0.002 (0.017) | -0.001 (0.020)

18. Secondary Outcome: Body Composition- Waist Circumference
Description: The annualized change in body composition measures over 3 years.
  Body composition slopes (trajectory over 3 years) were created for each participant with outcomes multiply imputed for children without body composition measurements post-baseline. An F test with two numerator degrees of freedom was used to test for between-group differences using an alpha of .05.
  Change in slope of waist circumference (cm) over time reported.
Time Frame: [Baseline, 12 mos, 24 mos, 36 mos]
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | HealthyCHANGE | SystemCHANGE | Tools4CHANGE
Number analyzed (Participants) | 109 | 114 | 114
cm/year | 1.814 (3.584) | 2.339 (2.839) | 2.200 (3.288)

19. Secondary Outcome: Body Composition- Percent Body Fat
Description: The annualized change in body composition measures over 3 years.
  Body composition slopes (trajectory over 3 years) were created for each participant with outcomes multiply imputed for children without body composition measurements post-baseline. An F test with two numerator degrees of freedom was used to test for between-group differences using an alpha of .05.
  Change in slope of body fat percentage over time reported. Body fat percentage calculated using Stevens equation.
Time Frame: [Baseline, 12 mos, 24 mos, 36 mos]
Measure: Mean (Standard Deviation); unit: percent/year
Arm/Group | HealthyCHANGE | SystemCHANGE | Tools4CHANGE
Number analyzed (Participants) | 109 | 114 | 114
percent/year | -0.246 (2.376) | 0.299 (1.889) | -0.044 (2.170)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | HealthyCHANGE | SystemCHANGE | Tools4CHANGE
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/123 | 0/119
Serious Adverse Events (participants affected / at risk) | 30/118 | 29/123 | 28/119
Other Adverse Events (participants affected / at risk) | 0/118 | 0/123 | 0/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HealthyCHANGE (N=118) | SystemCHANGE (N=123) | Tools4CHANGE (N=119)
Cardiac event (Cardiac disorders) | 4 (5) | 1 (1) | 3 (3) — Any event related to the cardiovascular system
Diabetic event (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) — Any event related to diabetes
Diabetes-related complications (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Surgery (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cancer diagnosis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hospitalization (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hospitalization (General disorders) | 4 (5) | 3 (3) | 4 (4)
Immune system disorder diagnosis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Immune system disorder complications (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Event resulting in injury or poisoning (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 2 (2) — Non-study related events only
Nervous system event (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Childbirth (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 3 (3) | 4 (4)
Pregnancy complications (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 2 (2)
Psychiatric event (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Event related to reproductive system (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0)
Respiratory event (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 3 (3)
Housefire (Social circumstances) | 0 (0) | 0 (0) | 2 (2)
Surgery (Surgical and medical procedures) | 7 (7) | 8 (8) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2012-03-30): https://cdn.clinicaltrials.gov/large-docs/79/NCT01514279/Prot_SAP_ICF_000.pdf